CLINICAL TRIAL: NCT04067284
Title: Does Early Initiation of Homemade Yogurt Supplementation Prevents Stunting - a Pilot Randomized Controlled Trial
Brief Title: Homemade Yogurt Supplementation to Prevent Stunting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Western Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-19062
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-08

CONDITIONS: Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A three-arm randomized controlled trial in Dhaka's slum area is proposed. Infants at risk of stunting (-1 SD length-for-age z-score, LAZ) aged around 5 months are eligible for the study. Eligible children will be randomised to receive: 1) nutrition education on dietary diversity; 2) a combination of similar education plus daily supplementation of homemade yogurt; 3) a 'usual care' (control) group. We will recruit 120 children (40 per arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education (Active Comparator): Nutrition education on dietary diversity.
  Interventions: Behavioral: Nutrition education
- Yogurt (Experimental): A combination of similar education plus daily supplementation of homemade yogurt
  Interventions: Dietary Supplement: Homemade yogurt supplementation
- Control (Active Comparator): Control group.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Nutrition education — Nutrition Education on
  * Continued breastfeeding until two years of age
  * Food groups
  * Balanced diet
  * Introduction to locally available nutritious and low-cost foods
  * Amount and frequency of complementary feeding
  * Safe water, and
  * Handwashing with soap before feeding
  Arms: Education
Dietary Supplement: Homemade yogurt supplementation — The homemade yogurt supplementation will start a week after beginning of 6 months of age once the child is introduced to solid foods of the mother's choice. The yogurt will be supplied to the mothers every day at time of feeding.
  Arms: Yogurt
Other: Usual care — No intervention/ control group
  Arms: Control

SUMMARY:
Stunting contributes substantially to child mortality and disease burden in low-income countries. In Bangladesh the prevalence of stunting among children <5-years of age is high (36%) reaching 50% in slum areas. The pathogenesis of stunting is multifaceted, yet nutritional inadequacy and repeated infections are established risk factors of stunting.

A three-arm randomized controlled trial in Dhaka's slum area is proposed. The children will be recruited from vaccination clinics. Infants at risk of stunting (-1 SD length-for-age z-score, LAZ) aged around 5 months are eligible for the study. Eligible children will be randomized to receive: 1) nutrition education on dietary diversity; 2) a combination of similar education plus daily supplementation of homemade yogurt; 3) a 'usual care' (control) group. The investigators will recruit 120 children (40 per arm). Intervention will be initiated a month before starting of complementary feeding with an educational session and will last 7 months during which a monthly educational session will be delivered at participant's household. The homemade yogurt supplementation will start a week after beginning of 6 months of age once the child is introduced to solid foods of the mother's choice. The yogurt will be supplied to the mothers every day at time of feeding. Feeding behaviors will be self-monitored using a pictorial calendar. Primary outcome (LAZ) and secondary outcomes (fecal bio-markers, WAZ, head circumference, and food diversity scores), will be measured at baseline (6 months), 9 months and 12 months of child age. Supplementation with homemade yogurt is a novel approach with the potential to improve infant gut environment, improve food absorption and thus potentially prevent stunting.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that, continued breastfeeding, adequate complimentary feeding and supplementation with homemade yogurt have the potential to reduce stunting.

Primary objective:

The present study is aimed to assess the impact of low-cost nutritional strategies to prevent childhood malnutrition in Bangladesh.

Specific objectives:

1. To compare differences in growth pattern (length-for-age z-score, weight-for age z-score, head circumference) of children at risk of stunting age 6-months between infants receiving educational program only, infants receiving education plus homemade yogurt supplementation and those receiving the "usual-care" (control).
2. To evaluate whether amount of gut microbiota necessary to improve gut health was associated with weight gain and growth in these children to support the casual mechanism behind this approach.

ELIGIBILITY:
Inclusion Criteria:

1. Infants at risk of developing stunting aged 5 months (-1SD LAZ)
2. All gender, religion, language and ethnicity
3. Infants born through normal delivery or cesarean section
4. Breastfeeding or non-breastfeeding

Exclusion Criteria:

1. Stunting or wasting (<-2SD LAZ)
2. Infants with any major congenital abnormality or any chronic conditions (e.g., rheumatic heart disease)

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline (6 months) length for age z-score (LAZ) at 9 months and 12 months of child age. | Will be measured at baseline (6 months), 9 months and 12 months of child age
  Child length converted to z-score

SECONDARY OUTCOMES:
Change from baseline (6 months) weight for age z-score (WAZ) at 9 months and 12 months of child age. | Will be measured at baseline (6 months), 9 months and 12 months of child age
  Child weight converted to z-score
Change from baseline (6 months) mean head circumference at 9 months and 12 months of child age. | Will be measured at baseline (6 months), 9 months and 12 months of child age
  Child head circumference
Change from baseline (6 months) mean concentration of fecal bio-markers at 9 months and 12 months of child age. | Will be measured at baseline (6 months), 9 months and 12 months of child age
  Concentration of neopterin, myeloperoxidase, and alpha 1 antitrypsin in stool samples.
Change from baseline (6 months) proportion of children meeting food diversity scores at 9 months and 12 months of child age. | Will be measured at baseline (6 months), 9 months and 12 months of child age
  * Minimum dietary diversity (MDD): the proportion of children who received foods from 4 or more food categories out of 7 specified categories on the previous day will be described as meeting the MDD score. Children will be divided into two groups, those who meet the above criteria will be scored 1 and those who do not meet the criteria will be scored 0.
  * Minimum meal frequency (MMF): the proportion of children who received solid, semi-solid, or soft foods the minimum numbers of time or more on the previous day will be described as meeting the MFF score. Children will be divided into two groups, those who meet the above criteria will be scored 1 and those who do not meet the criteria will be scored 0.
  * Minimum acceptable diet (MAD): the proportion of children who met both the MDD and MMF scores will be described as meeting the MAD score. MDD and MMF scores will be summed to estimate the MAD score. Children will be divided into two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Mahbubur Rahman, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided